CLINICAL TRIAL: NCT01886027
Title: Stress Management for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSU-022413B3E
Record Dates: First submitted 2013-06-13; First posted 2013-06-25 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Relaxation; Emotional exposure; Emotional Processing
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Emotional Awareness and Expression (Experimental): Emotional awareness and expression training (EAET) is an emotional processing intervention.
  Interventions: Behavioral: Emotional Awareness and Expression Training
- Relaxation (Active Comparator): Relaxation training will teach patients different relaxation training skills.
  Interventions: Behavioral: Relaxation Training
- Wait-list control (No Intervention): Standard medical care until the 3-month follow-up is completed

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Training — An emotional processing intervention, which aims to reduce stress by helping patients become aware of, and express emotions related to stressful life experiences, as well as teaching patients how to relate to others differently.
  Arms: Emotional Awareness and Expression
Behavioral: Relaxation Training — Teaches patients different relaxation training skills to reduce their distress and discomfort (i.e., progressive muscle relaxation, applied relaxation, or guided imagery.
  Arms: Relaxation

SUMMARY:
The primary goal of this study is to test the efficacy of emotional awareness and expression training (EAET), a novel emotional processing intervention that the investigators have developed, for people with IBS. In this randomized, controlled trial, the investigators will compare EAET to a standard intervention that teaches the conceptually opposite approach-relaxation training (RT)-and test how both of these interventions compare to a wait-list control condition. The investigators hypothesize that individuals in the EAET group will demonstrate greater improvement in their IBS symptom severity, psychological functioning, quality of life, and health care utilization at 4 and 12-week follow-up time points, compared to individuals in the wait-list control group. It is also expected that both of the active interventions (EAET and RT) will be more efficacious than the wait-list control condition.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate, individuals must meet the Rome III criteria for IBS. That is, they must report that they have had:

* recurrent abdominal pain or discomfort, or
* a change in stool frequency or form,
* at least three days per month, in the last three months, and
* that they have been given this diagnosis by a physician. They must also report having pain and discomfort of at least two days per week at time of screening.

Exclusion Criteria:

* Individuals who report having post-infectious IBS,
* organic gastrointestinal diseases (e.g., inflammatory bowel disease), immunodeficiency,
* a current psychotic disorder,
* drug or alcohol dependence within the past two years, and
* those who are unable to communicate in English will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
IBS symptom severity scale (IBS-SSS) | Change from baseline symptom severity at 1 month and 3 months

SECONDARY OUTCOMES:
McGill Pain Questionnaire, Short Form (SF-MPQ-2) | Change from baseline pain at 1 month and 3 months
Bristol Stool Form Scale (BSFS) | Change from baseline stool form at 1 month and 3 months
Irritable Bowel Syndrome, Quality of Life (IBS-QOL) | Change from baseline quality of life at 1 month and 3 months
Positive and Negative Affect Scale (PANAS) | Change from baseline positive affect and negative affect at 1 month and 3 months
Impact of Events Scale - Revised (IES-R) | Change from baseline impact of events at 1 month and 3 months
Toronto Alexithymia Scale -20 (TAS-20) | Change from baseline alexithymia at 1 month and 3 months
Rathus Assertiveness Schedule (RAS) | Change from baseline assertiveness at 1 month and 3 months
Ambivalence over Emotional Expression Scale (AEQ) | Change from baseline ambivalence over emotional expression at 1 month and 3 months
Emotional Approach Coping Scale (EAC) | Change from baseline emotional approach coping at 1 month and 3 months
IBS self-efficacy questionnaire | Change from baseline self-efficacy at 1 month and 3 months
Communicating Thoughts and Feelings Questionnaire | Change from baseline ability to communicate thoughts and feelings at 1 month and 3 months
Clinical Global Impressions (CGI) Improvement Scale - IBS version | Change from baseline IBS symptoms at 1 month and 3 months
Health care Utilization Scale | Change in health care utilization from baseline to 1-month and 3-month follow-ups
Brief Symptom Inventory | Change in psychological symptoms from baseline to 1-month and 3-month follow-ups
Early Trauma Inventory Self-Report Short Form | Change in Trauma reports from baseline to 1-month and 3-month follow-ups
Experiences in Close Relationships Questionnaire | Change in attachment from baseline to 1-month and3-month follow-ups
General Social Constraints Scale | Change in social constraints from baseline to 1-month and 3-month follow-ups
Medication use | Change in medication use from baseline to 1-month and 3-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Lumley, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Thakur ER, Holmes HJ, Lockhart NA, Carty JN, Ziadni MS, Doherty HK, Lackner JM, Schubiner H, Lumley MA. Emotional awareness and expression training improves irritable bowel syndrome: A randomized controlled trial. Neurogastroenterol Motil. 2017 Dec;29(12):10.1111/nmo.13143. doi: 10.1111/nmo.13143. Epub 2017 Jun 22. PMID 28643436